CLINICAL TRIAL: NCT05959226
Title: Effect of Exercise and Enteral Nutrition Intervention on Survival in Patients With Locally Advanced Gastric Cancer: a Prospective Multicenter Randomized Controlled Study
Brief Title: Effect of Exercise and Enteral Nutrition on Survival
Acronym: ENERGY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Quan Wang, Professor, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STARS-GC07
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Gastric Cancer; Nutrition Related Cancer; Sarcopenia
MeSH Terms: conditions — Stomach Neoplasms; Sarcopenia | interventions — Diet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise and Enteral Nutrition Intervention (Experimental): A comprehensive postoperative management combined physical exercise intervention with oral nutritional support
  Interventions: Behavioral: Exercise Intervention; Dietary Supplement: Nutrition Intervention
- Enteral Nutrition Intervention (Active Comparator): The control group will not receive exercise intervention, but will receive postoperative nutritional support treatment with the same standards as the experimental group.
  Interventions: Dietary Supplement: Nutrition Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — 1. Nutrition intervention: From discharge (7-14 days after surgery) until 6 months after surgery, patients are required to take 400 kcal/day of oral nutrition supplement (ONS) in addition to their normal diet..
  2. Exercise: under the guidance of the rehabilitation therapist, the patient gradually recovers Exercise from discharge (7-14 days after the operation) to 6 months after the operation, and should ensure at least 150 minutes of moderate intensity exercise or a combination of equivalent activities per week;
  Arms: Exercise and Enteral Nutrition Intervention
Dietary Supplement: Nutrition Intervention — (1) Nutrition intervention: From discharge (7-14 days after surgery) until 6 months after surgery, patients are required to take 400 kcal/day of oral nutrition supplement (ONS) in addition to their normal diet..

SUMMARY:
The present clinical trial was designed to explore the effect of postoperative physical exercise combined with enteral nutritional supplement on 3-year disease-free survival in patients with advanced gastric cancer.

DETAILED DESCRIPTION:
The present clinical trial was designed to explore the effect of physical exercise combined with enteral nutritional supplement on 3-year disease-free survival in patients with advanced gastric cancer. In the trial group, comprehensive postoperative management model with targeted exercise intervention and nutritional support. The details are as follows:

1. Nutrition intervention: From discharge (7-14 days after surgery) until 6 months after surgery, patients are required to take 400 kcal/day of enteral nutrition supplement (ONS) in addition to their normal diet. Once the patient's oral diet decreases, ONS will be added several times a day to ensure that the total energy reaches the ESPEN recommended daily 30 kcal/kg. The daily protein requirement is set at 1.2-1.5 g/kg of actual body weight. The Dietitian will keep records and help patients adjust their energy intake weekly.
2. Exercise: under the guidance of the rehabilitation therapist, the patient gradually recovers Exercise from discharge (7-14 days after the operation) to 6 months after the operation, and should ensure at least 150 minutes of moderate intensity exercise or a combination of equivalent activities per week; The control group patients received the same baseline evaluation as the experimental group patients. The control group will not receive phisical exercise intervention, but will receive postoperative nutritional treatment with the same standards as the experimental group.

ELIGIBILITY:
Inclusion Criteria:（1) 18 years ≤ age ≤ 70 years (2) Preoperative Karnofsky physical condition score: 0 or 1 or 2 (3) Preoperative pathological biopsy by gastroscope, histologically confirmed as adenocarcinoma (papillary adenocarcinoma, tubular adenocarcinoma, mucinous adenocarcinoma, Signet ring cell carcinoma, poorly differentiated adenocarcinoma, mixed adenocarcinoma) (4) Gastric cancer patients diagnosed with clinical stage Ib IIIc through CT, MRI, gastroscopy, and pathology (based on the 8th edition of UICC/AJCC staging) (5) Abdominal enhanced CT/MRI examination showed a clinical staging of cT2-4aN0-3M0 (based on AJCC-8thTNM tumor staging), and standard D2 radical surgery for gastric cancer was performed; (6) Have not received any radiotherapy, chemotherapy or immunotherapy; (7) Hemoglobin ≥ 80g/L; (8) Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; (9) Platelets ≥ 75 × 109/L; (10) ALT ≤ 2.5 times the normal upper limit value; (11) AST ≤ 2.5 times the normal upper limit value; (12) ALP ≤ 2.5 times the normal upper limit value; (13) Serum total bilirubin<1.5 times the upper normal limit value; (14) Serum creatinine<1 times the upper normal limit value; (15) Sign written informed consent;

Exclusion Criteria:

1. Patients diagnosed with distant metastasis through abdominal lung CT/MRI or PET-CT
2. Pregnant or lactating women
3. People with uncontrolled epilepsy, Central nervous system disease or mental disorders
4. Patients with combined limb disabilities or motor dysfunction;
5. Patients with other malignant diseases in the past five years, excluding cured skin cancer and cervical Carcinoma in situ
6. Clinically severe (i.e. active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) grade II or more severe congestive heart failure, or severe arrhythmia requiring medication intervention, or a history of myocardial infarction within the past 6 months
7. Have a history of cerebral infarction or cerebral hemorrhage in the past 6 months
8. Organ transplantation requires immunosuppressive therapy
9. Serious uncontrolled recurrent infections or other serious uncontrolled concomitant diseases
10. The patient has complications of Grade III or above in Clavien Dindo classification or has been hospitalized for more than 14 days after surgery due to various reasons;
11. Urgent surgery required due to tumor emergencies (bleeding, perforation, obstruction)
12. Pulmonary function test FEV1<expected value 50%
13. Received radiotherapy, chemotherapy, or other neoadjuvant treatment before surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival rate | 3 years after surgery
  The 3-year overall survival rate refers to the proportion of gastric cancer patients who have survived for more than 3 years after various comprehensive treatments

SECONDARY OUTCOMES:
3-year disease-free survival rate | 3 years after surgery
  The proportion of clinically confirmed complete remission to recurrence within 3 years
Scored Patient-Generated Subjective Global Assessment, PG-SGA | 6 months after surgery
  Scored Patient-Generated Subjective Global Assessment is the preferred method recommended by the American Dietitian Association for nutritional screening of tumor patients. It can conduct qualitative and quantitative comprehensive evaluation of patients' nutritional status from four aspects: weight loss, disease and age, metabolic stress status, and physical examination. It is a sensitive evaluation scale for patients to malnutrition changes
QLQ-C30 assessment | 6 months after surgery
  The quality of life of patients 6 months after surgery was evaluated using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30), which can evaluate the quality of life from a multidimensional perspective and better reflect the connotation of quality of life. It is widely used in clinical practice to measure the quality of life of cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Wang, Dr, Principal Investigator — The First Hospital of Jilin University

REFERENCES:
- [Background] Tegels JJ, van Vugt JL, Reisinger KW, Hulsewe KW, Hoofwijk AG, Derikx JP, Stoot JH. Sarcopenia is highly prevalent in patients undergoing surgery for gastric cancer but not associated with worse outcomes. J Surg Oncol. 2015 Sep;112(4):403-7. doi: 10.1002/jso.24015. Epub 2015 Aug 31. PMID 26331988
- [Background] Yu J, Huang C, Sun Y, Su X, Cao H, Hu J, Wang K, Suo J, Tao K, He X, Wei H, Ying M, Hu W, Du X, Hu Y, Liu H, Zheng C, Li P, Xie J, Liu F, Li Z, Zhao G, Yang K, Liu C, Li H, Chen P, Ji J, Li G; Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group. Effect of Laparoscopic vs Open Distal Gastrectomy on 3-Year Disease-Free Survival in Patients With Locally Advanced Gastric Cancer: The CLASS-01 Randomized Clinical Trial. JAMA. 2019 May 28;321(20):1983-1992. doi: 10.1001/jama.2019.5359. PMID 31135850
- [Background] Davis JL, Selby LV, Chou JF, Schattner M, Ilson DH, Capanu M, Brennan MF, Coit DG, Strong VE. Patterns and Predictors of Weight Loss After Gastrectomy for Cancer. Ann Surg Oncol. 2016 May;23(5):1639-45. doi: 10.1245/s10434-015-5065-3. Epub 2016 Jan 5. PMID 26732274
- [Background] Climent M, Munarriz M, Blazeby JM, Dorcaratto D, Ramon JM, Carrera MJ, Fontane L, Grande L, Pera M. Weight loss and quality of life in patients surviving 2 years after gastric cancer resection. Eur J Surg Oncol. 2017 Jul;43(7):1337-1343. doi: 10.1016/j.ejso.2017.01.239. Epub 2017 Feb 9. PMID 28222970
- [Background] Aoyama T, Sato T, Maezawa Y, Kano K, Hayashi T, Yamada T, Yukawa N, Oshima T, Rino Y, Masuda M, Ogata T, Cho H, Yoshikawa T. Postoperative weight loss leads to poor survival through poor S-1 efficacy in patients with stage II/III gastric cancer. Int J Clin Oncol. 2017 Jun;22(3):476-483. doi: 10.1007/s10147-017-1089-y. Epub 2017 Feb 7. PMID 28176023